CLINICAL TRIAL: NCT07006662
Title: Anatomical Landmarks for Chest Wall Perforators Used for Partial Breast Reconstruction (LaPBrecon)
Brief Title: Anatomical Landmarks for Chest Wall Perforators Used for Partial Breast Reconstruction
Acronym: (LaPBrecon)
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3427
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this 6-month proof-of-concept study is to map out the chest wall perforators in relation to anatomical landmarks for partial breast reconstruction.

DETAILED DESCRIPTION:
Breast conserving surgery is commonly performed in patients with breast cancer. It is important to fill the defect from a breast conserving procedure to achieve good cosmetic outcome. This defect can be filled either by using the adjacent breast tissue or by using perforator flaps; commonly taken from the area posterolateral to the breast or or below the inframammary crease. These perforator flaps can be based on thoracodorsal artery, lateral thoracic artery, lateral intercostal artery or the medial intercostal artery. The identification of these perforators using a hand-held doppler is an important but time-consuming intraoperative step. Surgeons often use the information derived from cadaveric studies when identifying these perforators as there is minimal information on the location of these perforators in relation to anatomical landmarks.

Patients with a BMI of < 25 Kg/m2admitted for elective breast surgery or attending breast outpatients' clinic will be included in the study. Patients will be sent information about this study prior to admission or the clinic appointment with a copy of the consent form. Participants will have a 30-minute assessment using a hand held doppler and perforators will be mapped against soft tissue and bony landmarks. Data will be analysed to identify common anatomical locations for the different chest wall perforators.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective breast surgery
* Age ≥ 18 years
* Female
* BMI ≤ 30 kg/m2
* Willing and able to give fully informed consent,
* Willing and able to comply with the study procedures

Exclusion Criteria:

* Pregnant patients
* Previous bilateral Breast or axillary surgery
* Undergoing bilateral oncoplastic procedure or requiring bilateral pre-operative marking
* Undergoing breast surgery requiring pre-operative marking of some of the landmarks and has had contralateral breast or axillary surgery in the past
* Surgery planned within 24 hours of screening for eligibility
* Known history of allergy or contact dermatitis to ultrasound gels

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The trial will be carried out at University Hospitals of North Midlands (UHNM). This will be a single centre study. Patients will be screened by the breast surgery Team for the eligibility criteria and recruited from the Breast Outpatients Clinic and marking of the perforators will be carried out on admission unit.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Location of vesselse | 6 months
  The location of the AICAP vessels in vertical and horizontal axis using constant bony and soft tissue landmarks. This will be measured by the distance of the perforators from the anatomical landmarks
Location of vessels | 6 months
  The location of the MICAP vessels in vertical and horizontal axis using constant bony and soft tissue landmarks. This will be measured by the distance of the perforators from the anatomical landmarks
Location of vessels | 6 months
  The location of the LTAP vessels in vertical and horizontal axis using constant bony and soft tissue landmarks. This will be measured by the distance of the perforators from the anatomical landmarks
Location of vessels | 6 months
  The location of the LICAP vessels in vertical and horizontal axis using constant bony and soft tissue landmarks. This will be measured by the distance of the perforators from the anatomical landmarks

SECONDARY OUTCOMES:
Variability | 6 months
  The degree of variability in location of the perforators.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom